CLINICAL TRIAL: NCT01861496
Title: Phase I/II Study to Evaluate the Safety and Tolerability of LiPlaCis (Liposomal Cisplatin Formulation) in Patients With Advanced or Refractory Tumours
Brief Title: Phase I/II Study to Evaluate the Safety and Tolerability of LiPlaCis in Patients With Advanced or Refractory Tumours
Acronym: LiPlaCis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Allarity Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LiPlaCis/P1/002; SMR-3338 (Other: Smerud Medical Research, Denmark)
Record Dates: First submitted 2013-05-01; First posted 2013-05-23 (Estimated); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Phase 1: Advanced or Refractory Solid Tumours; Phase 2 Part: Metastatic Breast Cancer, Prostate Cancer and Skin Cancer
Keywords: Cisplatin; Liposomal formulation; DRP (Drug Response Prediction)
MeSH Terms: conditions — Prostatic Neoplasms; Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LiPlaCis (Experimental): Dose escalation of LiPlaCis - a liposomal formulation of cisplatin will be administered intravenously in cycles every 3 weeks on day 1, day 8. Upon the investigator's judgement the patient may continue treatment for more than 3 cycles when benefiting from the study drug.
  Interventions: Drug: LiPlaCis

INTERVENTIONS:
Drug: LiPlaCis — LiPlaCis IV every 3 weeks on day 1, day 8
  Other Names: Liposomal formulation of Cisplatinum

SUMMARY:
Liposomal formulations are frequently used today in the treatment of cancer. LiPlaCis is the first targeted liposomal formulation with a tumour triggered release mechanism to undergo clinical development in oncology and it is expected that LiPlaCis will improve the therapeutic index of cisplatin compared to conventional cisplatin.

Cisplatin is one of the most widely used drugs in the treatment of cancer due to its documented efficacy in a number of tumour types. Furthermore, it seems highly likely that cisplatin will remain an important drug in the future treatment of cancer. However, the drug is associated with a number of serious toxicities that complicates or necessitates discontinuation of therapy - e.g. need for pre-hydration, neurotoxicity, nausea and vomiting.

Thus, there is a well-established need for improving cisplatin therapy in cancer patients. One option here is improving the formulation of the drug, so that a more selective up-take of cisplatin administered takes place at the tumour sites.

Based on the results of the pre-clinical studies of LiPlaCis, it seems clear that LiPlaCis offers the potential to improve cisplatin therapy to the benefits of cancer patients.

In a prematurely stopped Phase I Dutch study a Recommended Dose (RD) for a Phase II study was never reached which was the aim of the finished Phase I dose escalating part of this study for advanced or refractory solid tumors.

In the Phase 2 part of this study, patients with advanced breast cancer with a biopsy examination showing a pattern compatible with sensitivity to LiPlaCis or patients with skin cancer will be included.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological documented locally advanced or metastatic solid tumour relapsed on 2 or more different prior therapies. From step 5 and extension phase, population limited to Skin Cancer patients (non screened) or metastatic Breast Cancer patients or metastatic castration-resistant prostate cancer patients screened sensitive to LiPlaCis.
* Age >= 18 years.
* Life expectancy >= 3 months.
* ECOG performance status of 0 - 1.
* Recovered to Grade 1 or less from acute toxicities of prior treatment.
* >= 6 months must have elapsed since patient received cisplatin.
* >= 4 weeks must have elapsed since patient received any investigational medicinal product.
* >= 4 weeks must have elapsed since patient received any radiotherapy(except for palliative radiotherapy on non-target lesions), or treatment with cytotoxic or biologic agents (>=6 weeks for mitomycin or nitrosoureas). No hormonal treatment is allowed except treatment with corticosteroids at physiological dose and hormonal treatment with LHRH agonists for prostate cancer.
* >=2 weeks must have elapsed since any prior surgery or therapy with G-CSF and GM-CSF.
* Adequate condition as evidenced by the following clinical laboratory values:

  * Absolute neutrophil count (ANC) >= 1,5 x 10E9/L
  * Haemoglobin is at least 4,6 mmol/L
  * Platelets >= 75 x 10E9/L
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <= 2,5 x ULN, in case of known liver metastases ALT and AST <= 5 x ULN. Patients who does not conform to the transaminase inclusion criteria, but who by the PI are considered in good PS and otherwise eligible for inclusion, and where the transaminase levels are considered elevated due to other reasons than deteriorated liver capacity, may be considered for inclusion based on conferred agreement between PI and Sponsor
  * Serum bilirubin <= 1,5 ULN
  * Alkaline phosphatase <= 2,5 x ULN, in case of known liver metastases <= 5 x ULN. Patients who does not conform to the Alkaline phosphatase inclusion criteria, but who by the PI are considered in good PS and otherwise eligible for inclusion, and where the Alkaline phosphatase levels are considered elevated due to other reasons than deteriorated liver capacity, may be considered for inclusion based on conferred agreement between PI and Sponsor
  * Blood urea within normal limits, creatinine below upper normal limits and creatinine clearance within normal limits (>= 60 mL/min Cr-EDTA clearance).In the case of hydronephrosis, renography must be considered prior to treatment with LiPlaCis. For signs of drainage obstacle, well-functioning renal excretion/effect and normal diuresis must be ensured, e.g. via a double-J catheter.
* Sexually active males and females of child-producing potential, must use adequate contraception (oral contraceptives, intrauterine device or barrier method of contraception) for the study duration and at least six months afterwards.
* Patient must understand the investigational nature of this study and sign an independent ethical committee (IEC) approved written informed consent form prior to any study related activities.

Exclusion Criteria:

* Active uncontrolled bleeding or bleeding diathesis (e.g., active peptic ulcer disease).
* Any active infection requiring parenteral or oral antibiotic treatment.
* Known infection with human immunodeficiency virus (HIV) or hepatitis virus.
* Pre-existing renal insufficiency. Please refer to inclusion criteria no. 10g.
* Active heart disease including myocardial infarction or congestive heart failure within the previous 6 months, symptomatic coronary artery disease, or symptomatic arrhythmias currently requiring medication.
* Known or suspected active central nervous system (CNS metastasis). (Patients stable 8 weeks after completion of treatment for CNS metastasis are eligible).
* Autoimmune disease.
* Impending or symptomatic spinal cord compression or carcinomatous meningitis.
* Pre-existing neuropathy, i.e., Grade >1 neuromotor or neurosensory toxicity (as defined by National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) v4,0), except for abnormalities due to cancer.
* Known hypersensitivity to cisplatin or liposomes.
* Requiring immediate palliative treatment of any kind including surgery and/or radiotherapy(except for palliative radiotherapy on non-target lesions).
* Female patients who are pregnant or breast-feeding (pregnancy test with a positive result before study entry).
* Unwilling or unable to follow protocol requirements.
* Previous progression on a platinum containing therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-04; Primary Completion 2021-10 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and recommended dose (RD) by evaluating the safety and tolerability | one year
  Primary Objective:
  Assessment of adverse events and laboratory abnormalities

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentrations of platinum (Cmax) | Prior to the initial dose on day 1, day 8 and 15 and 5 min before end of infusion, 5 min, 0,5, 1, 3, 7, 24, 48, 72 hours post dose
  Blood samples are obtained and plasma concentrations of total LiPlaCis-derived platinum are determined using a validated atomic absorption spectrometry method.
Concentration of platinum (Pt-DNA) | Prior to the initial dose on day 1and 24 hours after
  Tumor and normal tissue biopsies are obtained concentrations of platinum are determined using a validated method.
Area Under the Plasma - Time Concentration Curve (AUC) | Prior to the initial dose on day 1, day 8 and 15 and 5 min before end of infusion, 5 min, 0,5, 1, 3, 7, 24, 48, 72 hours post dose
  Blood samples are obtained and plasma concentrations of total LiPlaCis-derived platinum are determined using a validated atomic absorption spectrometry method.
Elimination half-life of platinum (T½) | Prior to the initial dose on day 1, day 8 and 15 and 5 min before end of infusion, 5 min, 0,5, 1, 3, 7, 24, 48, 72 hours post dose
  Blood samples are obtained and plasma concentrations of total LiPlaCis-derived platinum are determined using a validated atomic absorption spectrometry method.
Total body clearance of platinum (Cl) | Prior to the initial dose on day 1, day 8 and 15 and 5 min before end of infusion, 5 min, 0,5, 1, 3, 7, 24, 48, 72 hours post dose
  Blood samples are obtained and plasma concentrations of total LiPlaCis-derived platinum are determined using a validated atomic absorption spectrometry method.
Volume of distribution of platinum at steady state (Vss) | Prior to the initial dose on day 1, day 8 and 15 and 5 min before end of infusion, 5 min, 0,5, 1, 3, 7, 24, 48, 72 hours post dose
  Blood samples are obtained and plasma concentrations of total LiPlaCis-derived platinum are determined using a validated atomic absorption spectrometry method.
Therapeutic efficacy of LiPlaCis (Efficacy Endpoint) | Tumor Assessed every 6 weeks until and at end of treatment, with an expected average of 3 treatment cycles (9 weeks)
  Response and progression is evaluated using internationally accepted response criteria and definitions proposed by the RECIST criteria.
Progression Free Survival | one year after end of treatment
  PFS for patients at dose step 5 and up by Response and progression evaluated using internationally accepted response criteria and definitions proposed by the RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Lassen, Professor MD, Ph.D, Principal Investigator — Rigshospitalet, Finsen Centre, Oncology Department, Phase 1 Unit; Dorte Nielsen, Professor MD, Ph.D, Principal Investigator — Herlev&Gentofte Hospital, Oncology Department
Locations (4):
- Denmark (4):
  - The Phase One Unit, The Finsen Centre, Rigshospitalet, Copenhagen
  - Herlev & Gentofte Hospital, Herlev
  - Nordsjællands Hospital Hillerød, Hillerød
  - Vejle Sygehus, Vejle